CLINICAL TRIAL: NCT04440787
Title: To Evaluate "Three Point Cuff Palpation Technique" for Assessing Optimal Depth of Endotracheal Tube Placement.
Brief Title: Prevention of Endotracheal Tube Migration by Cuff Palpation During Robotic Surgical Procedure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Amit Kumar Mittal, Consultant in-charge, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RES/SCM/30/2018/81
Record Dates: First submitted 2018-09-15; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Robotic Surgical Procedures
Keywords: Endotracheal intubation; pneumoperitoneum; trendelenburg position; Robotic surgery
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Three point cuff palpation and Blck mark line technique: In "Three point cuff palpation technique" the cuff will be palpated just below the cricothyroid membrane,at the level of suprasternal notch and below the suprasternal notchand the tube is re-positioned in case of any discrepancy between the black mark line technique and three point cuff at three different over the trachea.
  Interventions: Procedure: Three point cuff palpation technique

INTERVENTIONS:
Procedure: Three point cuff palpation technique — the ETT is finally positioned according to the Three point cuff technique.
  Other Names: Black line mark on the endotracheal tube

SUMMARY:
After intubation, the endotracheal tube was finally fixed after palpating endotracheal cuff at three sites (just below the cricoid cartilage, at suprasternal level and just below suprasternal notch). Fibre optic bronchoscopy will be done to find distance between tip of endotracheal tube and carina. This distance will be measured repeatedly, after pneumoperitoneum, after trendelenburg position and after making the patient supine at the end of surgery. Change in the distance will be noted.

DETAILED DESCRIPTION:
The endotracheal tube (ETT) will be placed according to the black mark on the tube, post-intubation, the tube will be finally fixed after palpating endotracheal cuff at three sites (below cricoid cartilage, at suprasternal level and just below suprasternal notch). ETT cuff position will be scanned by sonography of airway to confirm the position of the proximal end of the ETT cuff. Fibre optic bronchoscopy will be done to find distance between tip of endotracheal tube and carina. This distance will be measured repeatedly 5 minutes after pneumoperitoneum, 10 minutes after trendelenburg position and 10 minutes after making the patient supine at the end of surgery. Change in the distance will be noted to confirm the migration of ETT.

ELIGIBILITY:
Inclusion Criteria:

* Robotic uro-oncological surgical procedures of perineum
* Robotic gynae-oncological surgical procedures of perineum

Exclusion Criteria:

* Upper airway fibrosis or tracheal stenosis
* Large neck swelling distorting or deviating the trachea.
* Head and neck surgeries
* Laryngeal and tracheal tumour
* Tracheal surgery
* Previous tracheostomy
* previous radiation treatment of neck

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing the robotic urological or gynecological surgery in Trendelenburg position with pneumoperitoneum will be included in the study cohort.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-01-19 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Measure the distance between tip of endotracheal tube and Carina by fiber-optic bronchoscopy and measuring scale at various phases of robotic surgical procedure. | Throughout robotic surgical procedure, immediately after intubation, 5 minute after pneumoperitoneum, 10 minutes after trendelenburg position and after dedocking and making patient supine.pneumoperitoneum.
  proper endotracheal tube placement is labelled when the distance between the tip of tube and Carina is more than 2.5 cm, after placement the tube by three point cuff palpation technique, its position will be assessed at respective time points.

SECONDARY OUTCOMES:
find the effect of cricod cartilage and supra-sternal distance on endotracheal tube tip to Carina distance. | Throughout robotic surgical procedure, immediately after intubation, 5 minute after pneumoperitoneum, 10 minutes after trendelenburg position and after dedocking and making patient supine.
  cricoid cartilage to suprasternal distance changes with the position of neck, so it could affect the distance between the endotracheal tube tip and carina as the position of patient changes during various robotic surgical steps.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Kr Mittal, MD, Principal Investigator — Rajiv Gandhi Cancer Institute and Research centre
Locations (1):
- Rajiv Gandhi Cancer Institute & Research center, Rohini, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang CH, Lee HK, Nam SH. The displacement of the tracheal tube during robot-assisted radical prostatectomy. Eur J Anaesthesiol. 2010 May;27(5):478-80. doi: 10.1097/EJA.0b013e328333d587. PMID 19918180